CLINICAL TRIAL: NCT01865149
Title: Comparison of Optic Nerve Sheath Diameter on Retrobulbar Ultrasonography Before and After Drainage of Cerebrospinal Fluid in Pediatric Patient With Hydrocephalus
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 1-2013-0022
Record Dates: First submitted 2013-05-22; First posted 2013-05-30 (Estimated); Last update posted 2013-05-30 (Estimated); Status verified 2013-05

CONDITIONS: Hydrocephalus
Keywords: Child; Optic nerve sheath diameter; Hydrocephalus; Intracranial hypertension
MeSH Terms: conditions — Hydrocephalus; Intracranial Hypertension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- both optic nerve sheath diameter
  Interventions: Procedure: retrobulbar ultrasound

INTERVENTIONS:
Procedure: retrobulbar ultrasound — both optic nerve sheath diameter (the posterior 3mm of the papilla), 5 individual measurement

SUMMARY:
Studies in patients with intracranial hypertension have shown a good relationship between optic nerve sheath diameter measured by retrobulbar ultrasound and invasively measured intracranial pressure. The aim of this study was to evaluate changes in optic nerve sheath diameter before and after drainage of cerebrospinal fluid in patients with hydrocephalus.

ELIGIBILITY:
Inclusion Criteria:

1. ASA Ⅰ-Ⅱ
2. aged between 1 and 19 year
3. hydrocephalus
4. general anesthesia for undergoing drainage of cerebrospinal fluid

Exclusion Criteria:

1. an anatomical or functional abnormality in optic nerve

Ages: 1 Year to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: patient with hydrocephalus
Sampling Method: Non-Probability Sample
Enrollment: 38 (Estimated)
Dates: Start 2013-05; Primary Completion 2014-05 (Estimated); Study Completion 2014-05 (Estimated)

PRIMARY OUTCOMES:
both optic nerve sheath diameter (the posterior 3mm of the papilla) | For day 1 from induction of general anesthesia to average 15 min after recovery of general anesthesia

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Anesthesia and Pain Research Institute,, Seoul, Seoul, South Korea